CLINICAL TRIAL: NCT07302295
Title: Clinical and Socioeconomic Characteristics of Suicidal Behaviour in Children and Adolescents During the Covid19 Pandemic Period in Auvergne-Rhône-Alpes. Prospective Quantitative and Qualitative Study
Brief Title: Analysis of Suicidal Behavior Among Children and Adolescents in the Auvergne-Rhone-Alpes Region During the Covid 19 Pandemic Period
Acronym: TSPedCovid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL22_1175; 2023-A02237-38 (Other: ID-RCB)
Record Dates: First submitted 2025-11-24; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-11

CONDITIONS: Suicidality; COVID -19
Keywords: suicide; pediatrics; covid-19
MeSH Terms: conditions — Suicidal Ideation; COVID-19; Suicide | interventions — Data Collection

STUDY DESIGN:
Intervention Model Description: Multicenter descriptive study, involving retrospective data collection with a questionnaire and prospective qualitative evaluations. Research involving human subjects outside of health products as mentioned in Article L1121-1, 2° of the Public Health Code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects with suicidal behaviors during the health crisis of covid-19 between 2020 and 2022 (group1) (Experimental): * Name : Group 1
  * Subjects with Suicidal Behaviors (suicidal conduct, ideas, self-harm with suicidal intention) during the Health Crisis of Covid-19 and admitted to pediatric emergency services or hospitalized in a care unit (university hospital, general hospital) in the AURA region participating between 2020 and 2022.
  * Age ≥ 8 years old and < 18 years old between 2020 and 2022.
  Interventions: Other: Aggregated data collection
- Subjects with suicidal behaviors during covid-19 period with qualitative interviews (group 1b) (Experimental): * Name : Group 1b
  * Subjects with Suicidal Behaviors (suicidal conduct, ideas, self-harm with suicidal intention) during the Health Crisis of Covid-19 and admitted to pediatric emergency services or hospitalized in a care unit (university hospital, general hospital) in the AURA region participating between 2020 and 2022 and theirs parents
  * Age ≥ 8 years old and < 18 years old between 2020 and 2022 for subjects.
  * One or both parents
  * Subjects who agreed to participate in interviews and/or focus groups and gave their consent to be part of the group of patients participating in a qualitative interview (volunteer subjects).
  * Parent's subjects agreed their consent to be part of the group This group is estimated to 150 subjects and 300 parents max.
  Interventions: Other: Data collection and qualitative interview
- Subjects control with suicidal behaviors before the health crisis (Group 2). (Experimental): * Name: group 2
  * Subjects with suicidal behaviors (suicidal conduct, ideas, self-harm with suicidal intention) before the health crisis of Covid-19 (2018 and or 2019) and admitted to pediatric emergency services or hospitalized in a care unit (university hospital, general hospital) in the AURA region
  * Age ≥ 8 years old and < 18 years old between 2018 and 2019
  Interventions: Other: Aggregated data collection

INTERVENTIONS:
Other: Aggregated data collection — The demographic and diagnostic characteristics will be collected in aggregate form nafrom digital services departments or medical information departments of participating hospitals.
  Arms: Subjects control with suicidal behaviors before the health crisis (Group 2).; Subjects with suicidal behaviors during the health crisis of covid-19 between 2020 and 2022 (group1)
Other: Data collection and qualitative interview — The psychopathological and socioeconomic characteristics will be collected. For subjects who agreed, they will participate in interviews and/or focus groups. Parent's subjects who agreed will be part of focus groups too.
  Arms: Subjects with suicidal behaviors during covid-19 period with qualitative interviews (group 1b)

SUMMARY:
In 2020, the world is hit by a global health crisis due to a pandemic following the appearance of Sars-cov-2 or "covid-19". This pandemic was accompanied by a constant fear of contamination and death, relayed by the media. In France, the government proposed in response to the arrival of this virus on French territory. This policy was implemented in different ways over 3 distinct periods: strict containment at the start of the epidemic, then a "lighter" one, and finally a period of social restrictions without between these periods. This policy had a direct and rapid impact on the population's daily routines. Children and adolescents, are more susceptible to psychological trauma, as stress has a direct and psychic development. Studies have shown deleterious impact of the French health situation on the paediatric population. They point to an increase of psychological disorders such as depression and anxiety in the under -20s population, and an increase in suicidal gestures over the 2020-2021 period, with rates remaining higher than in previous years. Suicide is the 2nd leading cause of death in the population aged 15-24.

Studies continue to focus on the incidence of suicidal gestures of suicidal gestures and psychological disorders, and few of them examine the factors linked to the increase in these incidences, the traumatic impact or the story of the trajectory. Similarly, the few studies focus only on the population aged 12 and over, and in some cases, do not distinguish between age groups (15-24 or under 20).

Investigators believe that the various periods of social restrictions and eco-anxiety caused by the pandemic may have influenced suicidal behaviour in this population.

The main objective of this study is to investigate the clinical and socio-economic characteristics of the pediatric population who experienced suicidal behaviors in the Auvergne Rhone Alpes region during the covid 19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* The population (subjects and controls) will be divided into age categories:

  * Pre-adolescents (≥ 8 years and < 11 years)
  * Adolescents (≥ 11 years and < 15 years)
  * Older adolescents (≥ 15 years and < 18 years)

Subjects with suicidal behavior during the health crisis (Group 1):

* Age > 8 years and < 18 years during the period 2020 to 2022.
* Admitted to pediatric emergency departments or hospitalized in a care unit (CHU, general hospitals) in the AURA region during 2020, 2021, and/or 2022 for suicidal behavior (defined as suicidal ideation and/or suicide attempt and/or self-harm/self-poisoning with suicidal intent).

Subjects with suicidal behavior during the health crisis with qualitative interviews (Group 1b):

* Age > 8 years and < 18 years during the period 2020 to 2022.
* Admitted to pediatric emergency departments or hospitalized in a care unit (CHU, general hospitals) in the AURA region during 2020, 2021, and/or 2022 for suicidal behavior (defined as suicidal ideation and/or suicide attempt and/or self-harm/self-poisoning with suicidal intent).
* Randomly selected from the population of Group 1.
* For whom the parent(s) and/or the subject have signed informed consent.

Controls with suicidal behavior before the health crisis (Group 2):

* Age > 8 years and < 18 years during the period 2018 to 2019.
* Admitted to pediatric emergency departments or hospitalized in a care unit (CHU, general hospitals) in the AURA region during 2018 and/or 2019 for suicidal behavior (defined as suicidal ideation and/or suicide attempt and/or self-harm/self-poisoning with suicidal intent).

Exclusion Criteria:

- Subjects with Suicidal Behavior during the Health Crisis with and without Qualitative Interviews (Group 1 and 1b):

• Admitted to pediatric emergency services or hospitalized in a healthcare facility (university hospital center, general hospital) in the AURA region for a psychiatric reason other than suicidal behavior during the period from 2020 to 2022.

Controls with Suicidal Behavior before the Health Crisis (Group 2):

* Admitted to pediatric emergency services or hospitalized in a healthcare facility (university hospital center, general hospital) in the AURA region for a psychiatric reason other than suicidal behavior during the period from 2018 to 2019.
* Intercurrent illness with a life expectancy of less than 24 hours.

For Group 1:

* Pregnant, postpartum, or breastfeeding women.
* Persons deprived of liberty by judicial or administrative decision.
* Adults subject to a legal protection measure (guardianship, curatorship).
* Persons not affiliated with a social security scheme or beneficiaries of a similar scheme.
* Persons who do not understand and do not speak French.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6500 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Demographic and diagnostic characteristics | Baseline
  The following demographic and diagnostic characteristics will be collected in aggregate form for the entire population of children and adolescents who engaged in suicidal behavior during the health crisis and in the two preceding years:
  * Age, gender, place of residence,
  * ICD-10 diagnosis and referral,
  * Type of suicidal behavior (ideation, self-harm, suicide attempt),
  * Periods of social restrictions (lockdown, curfew, vaccine pass).

SECONDARY OUTCOMES:
Number of patients aged 8-17 and 11month admitted to pediatric emergency | Baseline
  Number of patients aged 8-17 and 11month admitted to pediatric emergency rooms or hospitalized in a continuous care/intensive care unit of university hospitals (CHU) or general hospitals (CH) for suicidal behavior during the COVID-19 pandemic period of 2020, 2021, and 2022, and those in the two preceding years: 2018 and 2019.
Psychopathological and socio-economic characteristics | Baseline
  The following psychopathological and socio-economic characteristics will be collected:
  * Age, sex, place of residence,
  * Family situation and intrafamilial relationships
  * Type of suicidal behavior and description (ideation, self-harm, suicide attempt)
  * Periods of social restrictions (lockdown, curfew, vaccination pass)
  * Leisure time and type of leisure activities/hobbies
  * Education
  * Relationship with peers
  * Previous and current psychiatric diagnosis (according to ICD-10)
  * Personal and family psychiatric history
  * Personal medical history
  * Pharmacological and psychological treatment; Type of care
Scores to CRIES | Up to 3 months
  Scores on the Children's Revised Impact of Events Scale (CRIES-13) (Horowitz et al., 1979; Brunet et al., 2003) among children from a representative sample of the cohort (group 1b, volunteer subjects).
CAS scale | Up to 3 months
  Scores on the Climate Anxiety Scale (CAS) (Clayton and Karazsia, 2020; Mouguiama-Daouda et al., 2022) among children from a representative sample of the cohort (group 1b, volunteer subjects).
Qualitative interview | Up to 3 months
  Semi-structured interviews with children and adolescents with suicidal behavior from a representative sample of the cohort.
  Subjects who agreed to interviews. We will try to have a sample of volunteers from Group 1 who can be representative of our population (care orientation, age, personal psychiatric history, and place of residence.)
Results to focus groups (parent's subjects, group 1b) | Up to 3 months
  Focus groups with the parents of children and adolescents with suicidal behavior from a representative sample of the cohort (randomly selected).

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hospices Civils de Lyon - Hôpital Femme Mère Enfant- Service de pédopsychiatrie de l'enfant et de l'adolescent, Bron
  - CHU de Clermont-Ferrand - Service de psychiatrie de l'enfant et de l'adolescent, Clermont-Ferrand
  - CHU de Grenoble - Service de psychiatrie de l'enfant et de l'adolescent, Grenoble
  - CHU de Saint-Etienne - Urgences psychiatriques, Saint-Etienne